CLINICAL TRIAL: NCT00177255
Title: A Phase II Study of Weekly Docetaxel (Taxotere®) in Combination With Capecitabine (Xeloda) in Advanced Gastric and Gastro-Esophageal Adenocarcinomas.
Brief Title: A Study of Docetaxel in Combination With Capecitabine in Stomach and Esophagus Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Roche has withdrawn support
Sponsor: University of Pittsburgh (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Nathan Bahary, MD, Associate Professor, Department of Medicine, Division of Oncology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-026
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: gastric; stomach; esophagus; esophageal
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel + Capecitabine (Experimental): Docetaxel 30mg/m2 will be administered as a 30-minute infusion on days 1 and 8. Each cycle will consist of 21 days. Premedication with dexamethasone will be given to all patients receiving weekly docetaxel therapy to reduce the incidence and severity of fluid retention as well as the severity of hypersensitivity reactions. Cycle 2 will begin on day 22.
  Capecitabine Capecitabine 825mg/m2 bid (total daily dose 1650mg/m2) will be administered orally for 14 days (days 1-14).
  Each cycle will consist of 21 days. Cycle 2 will begin on day 22.
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 30 mg/m2 will be administered as a 30-minute infusion on days 1 and 8. Each cycle will consist of 21 days.
  Cycle 2 will begin on day 22.
Drug: Capecitabine — Capecitabine 825 mg/m2 bid (total daily dose 1650 mg/m2) will be administered orally for 14 days (days 1-14).
  Each cycle will consist of 21 days.
  Cycle 2 will begin on day 22.
  Other Names: Capecitabine 825 mg/m2 bid (total daily dose 1650 mg/m2) will be administered orally for 14 days (days 1-14).; Each cycle will consist of 21 days.; Cycle 2 will begin on day 22.

SUMMARY:
This is a phase II study that will investigate weekly dosing of docetaxel in combination with capecitabine in advanced gastric and gastro-esophageal adenocarcinomas.

DETAILED DESCRIPTION:
This is a phase II study that will investigate weekly dosing of docetaxel in combination with capecitabine in advanced gastric and gastro-esophageal adenocarcinomas. Docetaxel 30mg/m2 will be administered on days 1 and 8 of each cycle and capecitabine 825mg/m2 bid (total daily dose 1650mg/m2) will be administered orally for 14 days (days 1-14) of each cycle. Each cycle is 21 days. Subjects will receive unlimited cycles of docetaxel and capecitabine until there is evidence of disease progression or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed locally advanced (unresectable) or metastatic adenocarcinoma of gastric, gastro-esophageal, or esophageal origin.
2. Must have measurable or evaluable disease.
3. Received adjuvant therapy are eligible if adjuvant therapy was given ≥ 6 months prior to the diagnosis of metastatic disease.
4. Life expectancy greater than 12 weeks.
5. ECOG performance status < 2.
6. Adequate organ and marrow function.
7. Preexisting peripheral neuropathy if present must be grade 0 or 1.
8. Women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 3 months thereafter. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential

Exclusion Criteria:

1. No chemotherapy or radiotherapy within 4 weeks
2. Not receiving any other investigational agents or participate in any investigational drug study within 4 weeks preceding the start of study treatment.
3. Patients with known brain metastases shall be excluded from this clinical trial
4. Patients with evidence or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant that precludes informed consent or interferes with the compliance of oral drug intake will also be excluded.
5. History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel, capecitabine or 5-FU.
7. Uncontrolled intercurrent illness
8. Pregnant or breast feeding women are excluded from this study
9. Inability to swallow tablets or those who have malabsorptive symptoms will be excluded.
10. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with docetaxel or capecitabine.
11. Prior use of docetaxel or capecitabine is not allowed ( Prior 5FU therapy is allowed).
12. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
13. Major surgery ( i.e laparotomy, line placement is not considered major surgery)within 4 weeks of the start of study treatment, without complete recovery.
14. Known, existing uncontrolled coagulopathy.
15. Patients on anticonvulsants that are metabolized via P450 3A4 pathway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahary, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel + Capecitabine: Docetaxel 30mg/m2 will be administered as a 30-minute infusion on days 1 and 8. Each cycle will consist of 21 days. Premedication with dexamethasone will be given to all patients receiving weekly docetaxel therapy to reduce the incidence and severity of fluid retention as well as the severity of hypersensitivity reactions. Cycle 2 will begin on day 22.
  Capecitabine Capecitabine 825mg/m2 bid (total daily dose 1650mg/m2) will be administered orally for 14 days (days 1-14).
  Each cycle will consist of 21 days. Cycle 2 will begin on day 22.
  Docetaxel: Docetaxel 30 mg/m2 will be administered as a 30-minute infusion on days 1 and 8. Each cycle will consist of 21 days.
  Cycle 2 will begin on day 22.
  Capecitabine: Capecitabine 825 mg/m2 bid (total daily dose 1650 mg/m2) will be administered orally for 14 days (days 1-14).
  Each cycle will consist of 21 days.
  Cycle 2 will begin on day 22.
Period: Overall Study
Arm/Group | Docetaxel + Capecitabine
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel + Capecitabine
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 61 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The time interval between the date on which a patient first received protocol treatment and the documented date of death.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel + Capecitabine
Number analyzed (Participants) | 39
Months | 10.7 [6.8 to 12.1]

2. Secondary Outcome: Overall Response Rate
Description: The number of responders (complete responders + partial responders) divided by the number of evaluable patients.
Time Frame: Every 2 cycles (6 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel + Capecitabine
Number analyzed (Participants) | 39
percentage of participants | 28.2 [15 to 44.9]

ADVERSE EVENTS:
Arm/Group | Docetaxel + Capecitabine
Serious Adverse Events (participants affected / at risk) | 20/39
Other Adverse Events (participants affected / at risk) | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Capecitabine (N=39)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Cardiovascular/General-Other (Cardiac disorders) | 2
Thrombosis/Embolism (Vascular disorders) | 1
Constitutional Symptoms-Other (General disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Ocular/Visual-Other (Eye disorders) | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Capecitabine (N=39)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 14
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 10
Constitutional Symptoms - Other (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 5
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5
Diarrhea (Gastrointestinal disorders) | 16
Dizziness (Nervous system disorders) | 4
Dry eye syndrome (Eye disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Edema: head and neck (General disorders) | 2
Edema: limb (General disorders) | 9
Edema: trunk/genital (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 26
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Flushing (Vascular disorders) | 4
Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 14
Hemorrhage, GI, Lower GI NOS (Gastrointestinal disorders) | 1
Hemorrhage, GI, Rectum (Gastrointestinal disorders) | 2
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 1
Injection site reaction/extravasation changes (General disorders) | 1
Insomnia (Psychiatric disorders) | 3
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1
Leukocytes (total WBC) (Investigations) | 5
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 2
Mood alteration, Depression (Psychiatric disorders) | 4
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 18
Nail changes (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 19
Neurology - Other (Nervous system disorders) | 10
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 12
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3
Ocular/Visual - Other (Eye disorders) | 1
Pain, Abdomen NOS (Gastrointestinal disorders) | 10
Pain, Anus (Gastrointestinal disorders) | 1
Pain, Back (Musculoskeletal and connective tissue disorders) | 7
Pain, Bone (Musculoskeletal and connective tissue disorders) | 1
Pain, Chest/thorax NOS (General disorders) | 2
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain, Head/headache (Nervous system disorders) | 1
Pain, Joint (Musculoskeletal and connective tissue disorders) | 1
Pain, Rectum (Gastrointestinal disorders) | 1
Pain, Stomach (Gastrointestinal disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelets (Investigations) | 3
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 17
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Rigors/chills (General disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 3
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Tremor (Nervous system disorders) | 1
Ulceration (General disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Vessel injury-vein, Other NOS (Injury, poisoning and procedural complications) | 1
Vision-blurred vision (Eye disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Watery eye (epiphora, tearing) (Eye disorders) | 7
Weight loss (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes